CLINICAL TRIAL: NCT06414187
Title: Clinical Effects of Intra-aortic Balloon Support in Early Acute Coronary Syndrome and Non-Acute Coronary Syndrome Related Cardiogenic Shock: a Multicenter Randomized Controlled Trial
Brief Title: Clinical Effects of Intra-aortic Balloon Support in Early Acute Coronary Syndrome and Non-Acute Coronary Syndrome Related Cardiogenic Shock
Acronym: IABP ON-TIME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Arrow International LCC (Subsidiary of Teleflex Inc.) (Unknown)
Responsible Party: Principal Investigator, Nicolas van Mieghem, Chair, Full Professional, Clinical Director of Interventional Cardiology, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IABP ON-TIME
Record Dates: First submitted 2024-01-03; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Cardiogenic Shock
Keywords: Intra-aortic balloon pump; Mechanical circulatory support; Acute coronary syndrome; Ischemic cardiogenic shock; Non-ischemic cardiogenic shock; Cardiogenic shock; Decompensated heart failure
MeSH Terms: conditions — Shock, Cardiogenic; Acute Coronary Syndrome | interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this trial will be 1:1 randomized to IABP support or standard of care (i.e. inotropes and/or vasopressors, but no IABP insertion). Patients will be stratified for ACS/non-ischemic etiology and stage B/stage C cardiogenic shock following stratification according to center.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Given the nature of percutaneous IABP support a double-blind trial design is not feasible. Therefore, this trial is an open-label randomized clinical trial indicating both the patient, treating physicians as well as researchers are aware of the allocated treatment (i.e. with or without IABP). The Clinical Event Committee (CEC), responsible for adjudicating events belonging to e.g. the primary outcome, are blinded for the allocated treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IABP-arm (Experimental): Patients assigned IABP therapy will undergo IABP insertion as promptly as possible, with a target interval from randomization to insertion of less than 30 minutes. Implantation of the IABP balloon can be established either in the cardiac catheterization laboratory or at bedside in the ICU or cardiac care unit. The steering committee of this trial recommends the use of an appropriate-sized IABP balloon according to the instructions for use.
  Low-dose vasopressors (noradrenaline/norepinephrine up to 0.2 ug/kg/min) are allowed next to IABP support. The necessity of increasing the noradrenaline/norepinephrine dose with at least 0.2 ug/kg/min or the necessity to initiate de-novo inotropic agents to reach a mean arterial blood pressure of at least 65 mmHg is considered treatment escalation.
  Interventions: Device: Intra-Aortic Balloon Pump
- Standard of care-arm (No Intervention): When a patient is randomized to the standard of care-arm, the definitive treatment strategy is up to the discretion of the treating physician (providing no IABP is inserted). The treatment strategy may include fluid management as well as administration of inotropes and vasopressors. The only imposed difference in treatment is the omission of IABP, as the dose of inotropes and vasopressors is not expected to be high in early cardiogenic shock.
  The final decision to escalate in the strategy of mechanical circulatory support (including to initiate IABP in the standard of care-arm) is up to the discretion of the treating physician. However, the steering committee feels escalation in MCS strategy is appropriate in case of persistent mean arterial pressure <65 mmHg with incessant lactate levels >5.0 mmol/L when pharmacologic support was already intensified (e.g. the noradrenaline/norepinephrine dose exceeds 0.2 ug/kg/min or inotropic support was already administered).

INTERVENTIONS:
Device: Intra-Aortic Balloon Pump — Patients who are randomized to the IABP-arm will be supported with IABP according to local, clinical guidelines (including algorithms for anticoagulation, verification of correct positioning and weaning strategies). The IABP console and disposables should be used according to the instructions for use, including the use of an appropriate-sized IABP balloon alligned with patient length and height.
  Arms: IABP-arm

SUMMARY:
The goal of this randomized controlled trial is to appraise the impact of intra-aortic balloon pump (IABP) in the treatment of early stages of cardiogenic shock, irrespective of etiology. Findings of this randomized trial may enhance clinical decision making regarding the use of MCS in specific subsets of patients in early stages of cardiogenic shock.

The main questions it aims to answer are:

* What are the effects of IABP on a composite of clinical endpoints representing clinical deterioration at 30-days in patients presenting with SCAI stage B or C cardiogenic shock?
* What is the 1-year clinical outcome (including mortality and hospital admissions for cardiovascular causes) of patients treated with vs. without IABP for early cardiogenic shock?
* Is there a difference in efficacy of IABP within the treatment of early cardiogenic shock related to Acute Coronary Syndrome versus non-ischemic causes?
* Is there a difference in efficacy of IABP within the treatment of SCAI stage B versus stage C cardiogenic shock?

Participants will be 1:1 randomized to IABP support or standard of care (a treatment strategy including inotropes and/or vasopressors but no IABP insertion). Patients will be stratified for Acute Coronary Syndrome/non-ischemic etiology and stage B/stage C cardiogenic shock, following stratification to center. Researchers will compare the group who was randomized to IABP to the control group (i.e. standard of care) to see if there is a difference in the primary trial endpoint after 30-days, including 1) all-cause mortality, 2) escalation to invasive mechanical ventilation, 3) escalation of mechanical circulatory support strategy, 4) acute kidney injury and 5) stroke or transient ischemic attack.

DETAILED DESCRIPTION:
Rationale: The scientific underpinning for the use of mechanical circulatory support (MCS) in early cardiogenic shock, especially for the intra-aortic balloon pump (IABP), is scarce and insufficiently clarified for different etiologies of cardiogenic shock. Previous randomized trials limited the inclusion criteria to patients with ischemic cardiogenic shock while observational research suggested favorable effects of timely adoption of IABP in patients with deteriorating myocardial function through ischemic or non-ischemic causes. Early stage of cardiogenic shock is defined by relative hypotension without hypoperfusion, or hypoperfusion still responsive to therapy (Society for Cardiovascular Angiography and Interventions, SCAI, stage B and C, respectively). A tightening of global guidelines with respect to the clinical adoption of IABP overshadowed the potential beneficial effects for specific patient categories within the total spectrum of cardiogenic shock. Patients currently presenting with early stages of cardiogenic shock caused by ischemic or non-ischemic etiology are hypothetically undertreated due to an assumed lack of clinical benefit of IABP in general. The aim of this randomized trial is to appraise the impact of IABP in the treatment of early stages of cardiogenic shock, irrespective of etiology. Findings of this randomized trial may enhance clinical decision making regarding the use of MCS in specific subsets of patients in early stages of cardiogenic shock.

Objective: The primary objective of this trial is to evaluate the 30-day clinical impact of IABP within the treatment of early (SCAI stage B or C) cardiogenic shock. Secondary objectives are

1) To evaluate the 1-year clinical outcome (including mortality and hospital admissions for cardiovascular causes) of patients treated with IABP for early cardiogenic shock; 2) To identify differences in efficacy of IABP in the treatment of early cardiogenic shock related to Acute Coronary Syndrome (ACS) versus non-ischemic causes; 3) To explore differences in efficacy of IABP in the treatment of stage B versus stage C cardiogenic shock.

Trial design: Open-label, multicenter, investigator-initiated, randomized controlled trial.

Trial population: The trial population consists of patients in early cardiogenic shock, defined as SCAI stage B or C, either related or unrelated to ACS.

Intervention: Patients enrolled in this trial will be 1:1 randomized to IABP support or standard of care (i.e. inotropes and/or vasopressors but no IABP insertion). Patients will be stratified for ACS/non-ischemic etiology and stage B/stage C cardiogenic shock following stratification according to center.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Stage B cardiogenic shock (presence of hypotension or tachycardia with signs of venous congestion, in absence of tissue hypoperfusion) OR
* Stage C cardiogenic shock (evidence of tissue hypoperfusion requiring any intervention beyond fluid management, still responsive to therapy) AND
* Must include at least one of the following: 1) lactate levels at least 2.0 mmol/L; 2) creatinine doubling OR >50 percent decline in glomerular filtration rate compared to baseline; 3) laboratory markers indicating liver injury (e.g. high serum transaminase levels) or 4) elevated NT-pro BNP.

A patient is eligible for trial inclusion if, at the time of randomization, no more than 1 inotropic agent has been administered AND when the maximum dose of noradrenaline/norepinephrine has not exceeded 0.2 ug/kg/min in the context of mean arterial pressure >65 mmHg.

Exclusion Criteria:

* The patient is in cardiogenic shock but does not fulfill the definition for stage B or C;
* Administration of at least 2 inotropic or vasopressive agents at study randomization;
* Administration of noradrenaline/norepinephrine exceeding 0.2 ug/kg/min at study randomization;
* Suspected or known mechanical complication contributing to cardiogenic shock, e.g. ventricular septal defect or papillary muscle rupture;
* Cardiogenic shock developing within 72 hours of a surgical procedure (i.e. low cardiac output with an inability to wean cardiopulmonary bypass);
* Inability to provide informed consent. Of not: patients admitted in cardiogenic shock who required cardiopulmonary resuscitation earlier, but are conscious at the time of hospital admission, are eligible for study participation;
* Known or suspected insufficiency of the aortic valve with at least moderate aortic regurgitation;
* Known or suspected peripheral arterial disease preventing safe insertion of IABP;
* Known or suspected thoracic or abdominal aortic disease (including aortic dissection or aortic aneurysm) precluding safe insertion of IABP;
* Suspicion of sepsis or septic shock (including septic cardiomyopathy);
* Pregnancy;
* Predicted life expectancy <6 months because of concomitant disease;
* Concurrent participation in a clinical trial with competing endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Composite primary endpoint (percent) | 30-days post enrollment
  The primary endpoint of the trial is the composite of the following outcomes: 1) all-cause mortality, 2) escalation to invasive mechanical ventilation, 3) escalation of mechanical circulatory support, 4) acute kidney injury and 5) stroke or transient ischemic attack.

SECONDARY OUTCOMES:
All-cause mortality (i.e. the individual determinants of the composite primary outcome) (percent) | 30-day follow-up
  See primary outcome (%) (based on details stated in patient's records)
Escalation to invasive mechanical ventilation (i.e. the individual determinants of the composite primary outcome | 30-day follow-up
  See primary outcome (%) (based on details stated in patient's records)
Escalation to mechanical circulatory support (i.e. the individual determinants of the composite primary outcome) | 30-day follow-up
  See primary outcome (%) (based on details stated in patient's records)
Acute kidney injury (i.e. the individual determinants of the primary outcome) | 30-day follow-up
  See primary outcome (%) (based on details stated in patient's records)
Stroke or transient ischemic attack (i.e. the individual determinants of the primary outcome) | 30-day follow-up
  See primary outcome (%) (based on details stated in patient's records)
Treatment escalation (percent) | 30-day follow-up
  Any steps in noradrenaline increase at least 0.2 ug/kg/min, or intensifying inotropic treatment (i.e. dose increasing or initiation of new agents) are considered treatment escalation, irrespective of trial arm. Uptitration of noradrenaline up to 0.2 ug/kg/min is considered standard of care. Treatment escalation also includes the initiation of MCS (including the institution of IABP in the standard of care-arm or escalation to e.g. continuous flow or extracorporeal mechanical circulatory support in the IABP-arm).
Deterioration of SCAI stage B to C (percent) | 30-day follow-up
  If the patient entered the trial meeting criteria for SCAI stage B
Deterioration of cardiogenic shock (percent) | at 7 and 14 days after randomization
  Degradation to SCAI stage D or E
Vascular complications defined according to VARC-3 guidelines (percent) | 30-day follow-up
  Following randomization to the IABP-arm, specifying major and minor vascular complications as well as major and minor access-related non-vascular complications
Major bleeding complications defined according to BARC guidelines (at least type 2) (percent) | 30-day follow-up
  Following randomization to the IABP-arm
De-novo Acute Coronary Syndrome (percent) | 30-day and 1-year follow-up
  i.e. type 1 myocardial infarction
Cardiopulmonary resuscitation or defibrillation (percent) | 30-day follow-up
  Including an appropriate shock of an Implantable Cardioverter Defibrillator
Development of SIRS, sepsis or severe sepsis (percent) | 96-hours after randomization
  Defined according to the Surviving Sepsis Guidelines

OTHER OUTCOMES:
Mortality (percent) | 30-day follow-up and 1-year follow-up
  Including presumed cause of death
Length of intensive care unit and hospital stay (in days) | 30-day follow-up
  Stay after randomization
Re-admission to the intensive care unit (percent) | 30-day follow-up
  After randomization
Implantation of Left Ventricular Assist Device or heart transplant (percent) | 30-day follow-up
  After randomization
Revascularization attempts (percent) | 30-day follow-up
  Including percutaneous coronary intervention or coronary artery bypass graft
1-Year composite endpoint (percent) | 1-year follow-up
  Including 1) all-cause mortality and 2) hospital admission because of cardiovascular disease
All-cause mortality (i.e. the individual determinants of the 1-year composite endpoint) | 1-year follow-up
  See 1-Year composite endpoint (percent), including 1) all-cause mortality and 2) hospital admission because of cardiovascular disease. Based on details stated in the patient's record.
Hospital admission because of cardiovascular disease (i.e. the individual determinants of the 1-year composite endpoint) | 1-year follow-up
  See 1-Year composite endpoint (percent), including 1) all-cause mortality and 2) hospital admission because of cardiovascular disease. Based on details stated in the patient's record.
Hospital re-admission (percent) | 1-year follow-up
  Including a description of the presumed cause of hospital (re-)admission
Visits to the emergency department (percent) | 1-year follow-up
  Of note, visits necessitating treatment escalation for heart failure
Unplanned revascularization (percent) | 1-year follow-up
  Including details concerning the revascularization attempt (i.e. percutaneous coronary intervention or coronary artery bypass graft)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas M Van Mieghem, Prof MD PhD, Study Chair — Erasmus Medical Center
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided